CLINICAL TRIAL: NCT00161031
Title: Atomoxetine as an Adjunct to Novel Antipsychotic Medication in the Treatment of Cognitive Deficits of Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, MPRC, PI, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-21702
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: Atomoxetine

SUMMARY:
The purpose of this study is to:

* To examine wether adjunctive atomoxetine is more effective thank placebo for neuropsychological measures of reaction time, motor speed, psychomotor speed, sustained attention, learning and memory, working memory, and executive functioning. To determine the effect size of atomoxetine on these neuropsychological measures for follow-up studies.
* To determine if atomoxetine has short-term benefits for improving weight gain and other metabolic abnormalities associated with antipsychotics.

DETAILED DESCRIPTION:
Participants with schizophrenia or schizoaffective disorder who are competent to participate in the informed consent process and provide written informed consent will be enrolled into the study. Participants will undergo a psychiatric evaluation, which will include the ascertainment of demographic information, past psychiatric and treatment history, and Structured Clinical Interview for DSM-IV (SCID; First et al, 1997) diagnostic interviews. A best estimate diagnostic approach will be utilized in which information from the SCID is supplemented by information from family informants, previous psychiatrists, and medical records to generate a diagnosis.

Clinical Assessments: The symptom assessments will include the Brief Psychiatric Rating Scale (BPRS; Overall and Gorham, 1961); Scale for the Assessment of Negative Symptoms (SANS; Andreasen, 1982); and Clinical Global Impression Scale (CGI; Guy, 1976). i) BPRS: the four positive symptom items - conceptual disorganization, suspiciousness, hallucinatory behavior, and unusual thought content - will be used to measure positive psychotic symptoms. These four items have been have been used to assess positive symptoms in previous studies (Kane et al, 1988; Buchanan et al, 1998). The BPRS Anxiety/Depression Factor, consisting of the somatic concern, anxiety, guilt feelings, and depression items, will be used to assess dysphoria (Guy, 1976). The BPRS hostility and uncooperativeness items will be used to assess hostility. We are not including the suspiciousness item, which is traditionally part of the BPRS Hostility Factor (Guy, 1976), because we have included this item with the other positive symptom items. ii) SANS: the SANS total score, minus the global items, inappropriate affect, poverty of content of speech, and attention items, will be used to measure negative symptoms. The inappropriate affect, poverty of content of speech, and attention items are excluded as lacking construct validity and because factor analytic study results suggest that these items are not closely related to negative symptoms (Buchanan and Carpenter, 1994). iii) CGI: the CGI severity of illness item will be used to assess global changes.

Safety Assessments: The safety assessments will include the Simpson-Angus Extrapyramidal Symptom Rating Scale (SAS; Simpson and Angus, 1970); Abnormal Involuntary Movement Scale (AIMS) (Guy, 1976); Barnes Akathisia Scale (BAS; Barnes, 1989) and Side Effect Checklist (SEC). i) SAS: a modified 11-item version of the SAS will be used to assess EPS. ii) AIMS: is a 12-item scale, with 7 items designed to assess abnormal facial, oral, extremity, and trunk movements; 3 global judgement items; and 2 current dental status items. iii) BAS : is a 4 item scale assessing objective and subjective symptoms of akathisia. iv) SEC: is designed to assess vital signs and commonly occurring antipsychotic side effects. v) Changes in total body weight, body mass index, lipid profile, and serum glucose.

Neurocognitive Assessments: The following neuropsychological tests will be administered: (1) reaction time, processing speed and efficiency, working memory-Digit Symbol, Number Sequencing, Letter Number Sequencing, Mental Arithmetic, Grooved Pegboard, Simple Reaction Time, Complex Reaction Time, Delayed Match to Sample from the Automated Neuropsychological Assessment Metric; (2) sustained attention and resistance to distractibility-Gordon's Continuous Performance Test; (3) learning and memory-California Verbal Learning Test and Brief Visual Memory Test; (4) executive functioning- Planning Test and Phonemic Fluency.

2-Week Stabilization Phase: In the 2-week stabilization phase, participants will undergo baseline symptom, medical, safety, and neurocognitive assessments. The participants will undergo a physical examination; an EKG; and laboratory tests of major organ functions (i.e., CBC, liver function tests, electrolytes, glucose, BUN/Creatinine, Urinanalysis (UA), and thyroid functions). A baseline antipsychotic level will be collected. All women will have a pregnancy test.

8-Week Double-Blind Treatment Phase: Participants will be randomly assigned to atomoxetine or placebo using a permuted block randomization system. Treatment assignment order is random within each block, and the total number of participants assigned to each treatment are equal. The block sizes will vary in random sequence between 2 and 4. Thus, it will be difficult to ascertain the next treatment assignment, even if a participant becomes unblinded, while the imbalance of numbers between the treatment groups is kept within tight limits. The central unblinded pharmacist will be notified of the treatment assignment, and will inform unblinded pharmacists at the other sites about which study medication to dispense. Separate emergency unblinding envelopes for each participant will be kept in a locked cabinet at each dispensing pharmacy. In addition, an emergency unblinding tool will allow specific, designated staff (i.e., the P.I. and Co-P.I.) to log onto the randomization data base through the MPRC computer network and request treatment assignment for a specific participant. An electronic audit trail will be kept of all such unblinding requests. All unused unblinding envelopes must be returned unopened to the central pharmacy at the end of the study. Participants will receive biweekly BPRS, SANS, SAS, BAS, AIMS, Side effect, and vital sign assessments. Neurocognitive assessments will be performed at week 0 and week 8 or endpoint. Laboratory tests, antipsychotic levels, and the EKG will be repeated at 8 weeks.

Medication Titration Schedule: The target atomoxetine dose for this study is 80 mg/day. The following titration schedule will be used: Week 1-2: atomoxetine 40 mg/day; Week 3-8: atomoxetine 80 mg/day. This titration schedule serves to enhance tolerability and minimize side effects. Participants randomized to placebo will receive an equal number of placebo tablets during the titration schedule.

Concomitant Medications: Participants in the study will be allowed to continue on their medication regimen that they were taking prior to the trial. This will allow the results to be more generalizable. Patients must be stabilized on a single second generation antipsychotic, excluding clozapine, at an unchanged dose for at least 4 weeks prior to randomization. All participants must be on a stable dose of all other psychotropic medications for at least 4 weeks prior to randomization. No medication changes or changes in dose will be permitted during the study period.

Because of atomoxetine's noradrenergic activity and it's modest ability to cause increases in blood pressure, participants on drugs that have the potential for vasopressor effects, such as venlafaxine or monoamine oxidase inhibitors, will be excluded.

Participants will be allowed as needed (PRN) benztropine (1-6mg/day) for extrapyrmidal symptoms, lorazepam (1-6 mg/day) for anxiety, agitation or akathisia, and chloral hydrate for sleep (500-1000 mg/day). To minimize the effects of the PRN medications on test results, participants will not receive any of the above PRN medications 12 hours prior to neurocognitive testing. Additionally, participants requesting the use of benztopine or any antiparkinson agent will first be assessed with a movement rating scale to document the presence of EPS prior to receiving the antiparkinson agent and will not have received any antiparkinson agent within 12 hours prior to the movement assessment. Participants requiring routine use of benztropine and lorazepam will be excluded or withdrawn from the study.

Maintenance of the Blind: For outpatients, study medication will be dispensed on a biweekly basis. They will be given two extra days of medication in case of a missed appointment. Inpatient subjects will receive their study medication daily from either the Spring Grove Hospital Center TRU or the Perry Point VAMHC central pharmacy. An unblinded pharmacist at each site will dispense all study medications. The blind will be broken only if a medical emergency requires this information. If this occurs, the participant will be withdrawn from the study.

All raters, investigators and other staff will be blind to treatment assignment except for the pharmacist. The pharmacist does not participate in assessing any of the primary symptom or side effect dependent variables and conveys no information about treatment assignment to participants or staff except in a medical emergency.

Compliance: Participants receiving 75% of their assigned medication will be considered compliant. The 75% criterion ensures that participants will receive adequate treatment to evaluate the comparative efficacy of atomoxetine and placebo. Outpatient compliance will be monitored through weekly pill counts and subject interviews. Medications will be dispensed on a weekly basis and will only be dispensed after compliance is assessed and all assessments are completed. Inpatient compliance will be monitored through inpatient medication records. If a participant is observed to have a compliance problem, then this will be discussed with the participant and a plan formulated to bring the participant back within the compliance parameter. For outpatients, the plan may include contacting the participant's caretaker or scheduling increased clinic visits. These monitoring procedures have been used in other MPRC studies and have resulted in high levels of compliance. Compliance patterns will be carefully monitored in each treatment group and will be described as part of any presentation of study results.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of either schizophrenia or schizoaffective disorder.
* Caucasian or Non-Caucasian.
* Subjects will be currently treated with one of the new generation antipsychotics: olanzapine, risperidone, quetiapine, or ziprasidone.
* Subjects will meet a prior criteria for cognitive impairment severity. The RBANS will be used to determine the level of cognitive impairment.

Exclusion Criteria:

* History of an organic brain disease.
* History of DSM-IV alcohol or substance abuse (within the last month), or DSM-IV alcohol or substance dependence (within the last six months).
* Pregnant women.
* Uncontrolled hypertension defined as high blood pressure exceeding 140/90 on three consecutive readings despite adequate treatment.
* Subjects receiving venlafaxine.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-04 (Actual); Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Is adjunctive atomoxetine is more effective than placebo for neuropsychological measures of reaction time, motor speed, psychomotor speed, sustained attention, learning and memory, working memory, and executive function.

SECONDARY OUTCOMES:
Examine whether adjunctive atomoxetine is more effective than placebo for positive symptoms and negative symptom measures.

CONTACTS AND LOCATIONS:
Overall Officials: Deanna L Kelly, Pharm.D., Principal Investigator — MPRC
Locations (2):
- United States (2):
  - Veterans Affairs Maryland Health Care System, Baltimore, Maryland
  - Maryland Psychiatric Research Center, Catonsville, Maryland

REFERENCES:
- [Derived] Kelly DL, Buchanan RW, Boggs DL, McMahon RP, Dickinson D, Nelson M, Gold JM, Ball MP, Feldman S, Liu F, Conley RR. A randomized double-blind trial of atomoxetine for cognitive impairments in 32 people with schizophrenia. J Clin Psychiatry. 2009 Apr;70(4):518-25. doi: 10.4088/jcp.08m04358. Epub 2009 Apr 7. PMID 19358788